CLINICAL TRIAL: NCT06292130
Title: FHIR-ed Up for Tobacco Cessation: Health-Kit Enabled Mobile App for Tobacco Cessation
Brief Title: Health-Kit Enabled Mobile App for Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sara Johnson, Co-President & CEO, Pro-Change Behavior Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156588-01; 1R43HL156588-01A1 (NIH)
Record Dates: First submitted 2022-02-28; First posted 2024-03-04 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cigarette Smoking
Keywords: smoking; app
MeSH Terms: conditions — Cigarette Smoking; Smoking; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single group, repeated measures (2 timepoints)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App users (Experimental): All participants will be provided with access to the intervention app (refresh).
  Interventions: Behavioral: refresh

INTERVENTIONS:
Behavioral: refresh — A theoretically-grounded, highly individualized tobacco cessation Health-Kit enabled app. Unlike existing tobacco cessation apps, refresh: 1) implements a full range of best practices in tailored health behavior change communications; 2) individualizes messaging based on the patient's clinical context using Health app data obtained through Fast Healthcare Interoperability Resources (FHIR) standard Application Programming Interfaces (API) and behavior change constructs; and 3) provides data and key insights back to the EHR.

SUMMARY:
Tobacco use is the leading preventable cause of death in the US, contributing to more than 480,000 premature deaths each year. The Tobacco Treatment Guidelines underscore the need to offer patients who use tobacco products brief interventions that include prescriptions for proven pharmacological smoking cessation aids and proactive connections to evidence-based behavioral support. The rapid expansion of smart phone capabilities enhances the potential for tobacco cessation apps to personalize behavior change guidance and to send contextually relevant tailored behavior change nudges based on readiness to quit and electronic heath record (EHR) data. Rich data from EHRs are now available to third-party apps from the Health app (iOS) via Fast Healthcare Interoperability Resources standard Application Programming Interface (API).

This Phase I Small Business Innovation Research (SBIR) explored the effects of one such innovative health IT solution. refresh is a highly individualized tobacco cessation HealthKit enabled app that 1) implemented a full range of best practices in tailored health behavior change communications based on readiness to change; 2) provided individualized behavior change guidance based on Health app data; and 3) concisely provided data and documentation of key actionable insights in the EHR on the patient's smoking status, app usage, and brief micro-message delivered by clinicians to reinforce and accelerate a patient's behavior change progress. This interoperability provided value to both patients and clinicians; empowered and supported successful and lasting behavior change; and enabled the implementation and evaluation of a best-in-class approach to tobacco and nicotine treatment.

Extensive end user and stakeholder input ensured that refresh was designed for rapid dissemination. Patients of an integrated delivery system with an upcoming appointment (n=51) were recruited to participate in a 30-day pilot test. Pre-post comparisons of Patient-Reported Outcomes Measurement Information System (PROMIS) measure for tobacco (psychosocial expectancies) and confidence for quitting provided preliminary data on the effects of the program. The hypothesis was that the patients who utilize refresh will have significantly higher psychosocial expectancies regarding tobacco at follow-up and greater confidence to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current cigarette smoker
* Having an iPhone 6s or higher
* Willing and able to download a mobile app
* Able to read and speak English
* Having an upcoming appointment with a participating clinician in the next 42 days

Exclusion Criteria:

* Younger than 18
* Non-smoker
* Unable to read and speak English
* Not having an iPhone 6s or higher
* Not having an appointment with a participating clinician in the next 42 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Johnson, Ph.D., Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (1):
- Pro-Change Behavior Systems, Inc, South Kingstown, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
A variety of peer-reviewed publications will emerge from the proposed research. At the conclusion of the study, the data will be de-identified and then made available to those requesting access, provided that they sign an agreement that the data will be used for research purposes only. Pro-Change routinely asks those requesting access to any data to sign such a form.

RESULTS

PARTICIPANT FLOW:
Groups:
- App Users: All participants will be provided with access to the intervention app (refresh).
  refresh: A theoretically-grounded, highly individualized tobacco cessation Health-Kit enabled app. Unlike existing tobacco cessation apps, refresh: 1) implements a full range of best practices in tailored health behavior change communications; 2) individualizes messaging based on the patient's clinical context using Health app data obtained through Fast Healthcare Interoperability Resources (FHIR) standard Application Programming Interfaces (API) and behavior change constructs; and 3) provides data and key insights back to the electronic health record (EHR).
Period: Overall Study
Arm/Group | App Users
Started | 51
Completed | 39
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | App Users
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 18
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Psychosocial Expectancies (PROMIS Smoking Initiative) Patient Reported Outcome
Description: This reliable and valid 6-item assessment measures feelings of social disapproval of smoking, normative values associated with smoking, and negative beliefs about appearance when smoking (e.g., If I quit smoking I will be more in control of my life). It will be the primary outcome as it is appropriate for all smokers (ready to quit or not) and is highly correlated with interest in quitting (r=0.59). It is also correlated with recency of quit attempts. Participants respond on a 5-point Likert Scale from 0 (Not at all) to 4 (Very much). Raw scores range from a minimum of 0 to a maximum of 24, with higher scores indicating better outcomes. The reliability of the scale is 0.85.
Time Frame: Pretest (baseline) and Posttest (30 day follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App Users
Number analyzed (Participants) | 39
score on a scale
  Pretest (baseline) | 12.7 (6.8)
  Posttest (30 day follow-up) | 13.6 (5.6)
Statistical Analysis 1: Comparison: App Users; Test type: Other; p = 0.17, t-test, 2 sided

2. Secondary Outcome: Confidence
Description: This 3-item scale assesses an individual's confidence level to refrain from using tobacco even in difficult situations and is a leading indicator of movement to cessation. Ratings of confidence will be made on a 5-point Likert scale (1=not at all; 5=extremely confident). Raw scores range from a minimum of 3 to a maximum of 15, with higher scores indicating better outcomes.
Time Frame: Pretest (baseline) and Posttest (30 day follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App Users
Number analyzed (Participants) | 39
score on a scale
  Pretest (baseline) | 6.3 (2.5)
  Posttest (30 day follow-up) | 7.6 (2.7)
Statistical Analysis 1: Comparison: App Users; Test type: Other; p = 0.006, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- App Users: All participants were provided with access to the intervention app (refresh).
  refresh: A theoretically-grounded, highly individualized tobacco cessation Health-Kit enabled app. Unlike existing tobacco cessation apps, refresh: 1) implements a full range of best practices in tailored health behavior change communications; 2) individualizes messaging based on the patient's clinical context using Health app data obtained through Fast Healthcare Interoperability Resources (FHIR) standard Application Programming Interfaces (API) and behavior change constructs; and 3) provides data and key insights back to the EHR.
Arm/Group | App Users
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT06292130/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT06292130/SAP_001.pdf
  • Informed Consent Form (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT06292130/ICF_002.pdf